CLINICAL TRIAL: NCT00723892
Title: Observatory on Treatment Adhesion in Patients Suffering From Hepatitis C Chronic Treated With ViraferonPeg® Injected / Rebetol® in Conjunction With a Psychotherapeutic Assistance Program
Brief Title: Adherence in Patients Receiving PegIntron/Rebetol for Hepatitis C in Conjunction With a Psychotherapy Support Program (Study P04252)
Status: Completed | Type: Observational
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: P04252; MK-4031-245 (Other: Merck)
Record Dates: First submitted 2008-07-25; First posted 2008-07-29 (Estimated); Results first posted 2010-09-20 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Hepatitis C, Chronic; Hepacivirus
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- PegIntron/Rebetol and psychotherapy support program: Participants receiving a psychotherapy support program during PegIntron/Rebetol therapy for hepatitis C.
  Interventions: Biological: Peginterferon alfa-2b (PegIntron); Drug: Rebetol (Ribavirin); Behavioral: Psychotherapy support program
- PegIntron/Rebetol alone (no psychotherapy): Participants receiving no psychotherapy support program during PegIntron/Rebetol therapy for hepatitis C.
  Interventions: Biological: Peginterferon alfa-2b (PegIntron); Drug: Rebetol (Ribavirin)

INTERVENTIONS:
Biological: Peginterferon alfa-2b (PegIntron) — Peginterferon alfa-2b (PegIntron) was administered based on the prescribed dose. The average dose for PegIntron was a weekly injection of 1.5 ± 0.3 μg^kg^week
  Other Names: PegIntron pen; SCH 54031; ViraferonPeg
Drug: Rebetol (Ribavirin) — Rebetol was administered orally based on the prescribed dose. The average dose for Rebetol was 950 ± 167.2 mg^day
  Other Names: Ribavirin; SCH 18908
Behavioral: Psychotherapy support program — Each site has implemented a psychotherapy support program.
  Groups: PegIntron/Rebetol and psychotherapy support program

SUMMARY:
Several psychiatric adverse events (eg, depression, fatigue, psychoses, behavior troubles, anxiety, irritability, deteriorated concentration, and insomnia) that are likely to occur during the treatment course with PegIntron plus Rebetol may prompt patients to discontinue their treatment early. The goal of this study is to assess whether a psychotherapy support program may contribute to a better adherence rate.

DETAILED DESCRIPTION:
Enrollment of participants will occur in a sequential order of treatment initiation.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with hepatitis C

Exclusion Criteria:

* According to the products' labeling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants at sites in France who are receiving a psychotherapy support program during therapy for hepatitis C and a control group without a psychotherapy support program.
Sampling Method: Probability Sample
Enrollment: 614 (Actual)
Dates: Start 2005-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 614 participants were recruited in this study.
Pre-assignment Details: Only 568 participants were assigned to treatment as they were foreseen to complete treatment, were consulted, and met inclusion criteria.
Period: Overall Study
Arm/Group | PegIntron/Rebetol and Psychotherapy Support Program | PegIntron/Rebetol Alone (no Psychotherapy)
Started | 313 | 255
Completed | 206 | 168
Not Completed | 107 | 87
Not completed — Participant not tracked | 33 | 35
Not completed — Virological criterion | 24 | 9
Not completed — Withdrawal by Subject | 6 | 9
Not completed — End planned | 11 | 7
Not completed — Bad tolerance | 5 | 5
Not completed — Multiple reasons | 17 | 12
Not completed — Other | 6 | 3
Not completed — Study end | 1 | 3
Not completed — Weight loss | 1 | 3
Not completed — Alcohol abuse | 0 | 1
Not completed — Intercurrent infection | 2 | 0
Not completed — Drug addiction | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PegIntron/Rebetol and Psychotherapy Support Program | PegIntron/Rebetol Alone (no Psychotherapy) | Total
Number analyzed (Participants) | 313 | 255 | 568
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants foreseen to complete treatment, consulted and assigned to treatment were analyzed.
  years | 45.5 (10.7) | 48.5 (11.8) | 46.8 (11.3)
Sex/Gender, Customized [Number; unit: participants] — Participants foreseen to complete treatment, consulted and assigned to treatment were analyzed.
  participants
    Female | 117 | 80 | 197
    Male | 195 | 175 | 370
    Unavailable (missing data) | 1 | 0 | 1
Region of Enrollment [Number; unit: participants] — Participants foreseen to complete treatment, consulted and assigned to treatment were analyzed.
  participants
    France | 313 | 255 | 568

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Complete Treatment With PegIntron/Rebetol Therapy for Hepatitis C When Administered With a Patient Psychotherapy Support Program as Compared to a Group Without a Psychotherapy Support Program.
Time Frame: 12 months after onset of treatment
Population: Participants foreseen to complete treatment, consulted and assigned to treatment were analyzed.
Measure: Number; unit: Participants
Arm/Group | PegIntron/Rebetol and Psychotherapy Support Program | PegIntron/Rebetol Alone (no Psychotherapy)
Number analyzed (Participants) | 313 | 255
Participants | 206 | 168

2. Secondary Outcome: the Average Length of Treatment for Participants on Treatment for Hepatitis C With PegIntron Pen/Rebetol
Time Frame: 12 months after onset of treatment
Population: Participants with no missing results.
Measure: Mean (Standard Deviation); unit: Weeks
Groups:
- PegIntron/Rebetol Alone (no Psychotherapy: Participants receiving no psychotherapy support program during PegIntron/Rebetol therapy for hepatitis C.
Arm/Group | PegIntron/Rebetol and Psychotherapy Support Program | PegIntron/Rebetol Alone (no Psychotherapy
Number analyzed (Participants) | 306 | 252
Weeks | 36.1 (16.2) | 35.3 (17.3)

ADVERSE EVENTS:
Description: Adverse events and serious adverse events were based on the number of participants recruited and enrolled (N=614).
Arm/Group | All Enrolled Participants
Serious Adverse Events (participants affected / at risk) | 11/614
Other Adverse Events (participants affected / at risk) | 0/614
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Enrolled Participants (N=614)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 1 (1)
Basedow's Disease (Endocrine disorders) | 1 (1)
Drug Intolerance (General disorders) | 1 (1)
Bronchopulmonary Aspergillosis (Infections and infestations) | 1 (1)
Pulmonary Tuberculosis (Infections and infestations) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Transient Ischemic Attack (Nervous system disorders) | 1 (2)
Persecutory Delusion (Psychiatric disorders) | 1 (1)
Dermatitis Exfoliative (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Data publishing of the observational study is forbidden. Data and results of the observational study are the exclusive property of the Sponsor.